CLINICAL TRIAL: NCT05773547
Title: Investigation of the Learning Effect in the Measurement of Circulation in Calf Muscle Using the Multispectral Optoacoustic Tomography
Brief Title: Investigation of the Learning Effect in the Measurement of Circulation in Calf Muscle Using MSOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Other Study IDs: MSOT_Lerneffekt
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Multispectral Optoacoustic Tomography; Learning Curve; Image Interpretation, Computer-Assisted; Structural Similarity Index Measure
Keywords: Multispectral Optoacoustic Tomography; Learning Curve; Learning Effect; MSOT; Image Interpretation; Structural Similarity Index Measure; SSIM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Professional: Two investigators who have performed over 200 MSOT measurements.
  Interventions: Device: MSOT measurements
- Trainee-personal teaching: Trainees are defined as who haven't performed any MSOT measurement. In this cohort, one trainee received a personal teaching from one professional.
  Interventions: Device: MSOT measurements
- Trainee-video: Trainees are defined as who haven't performed any MSOT measurement. In this cohort, one trainee received instruction from video.
  Interventions: Device: MSOT measurements
- Trainee-instruction in paperform: Trainees are defined as who haven't performed any MSOT measurement. In this cohort, one trainee received instruction in paperform.
  Interventions: Device: MSOT measurements

INTERVENTIONS:
Device: MSOT measurements — Non-invasive transcutaneous imaging of subcellular muscle components via infrared and near-infrared laser pulses

SUMMARY:
The goal of this observational study is to investigate the learning effect in the measurement of micro-circulation in healthy participants using MSOT. The main question it aims to answer are:

If there if a learning effect in MSOT measurement. How long does it takes for the trainees to reach the professional level. Is there a difference between different learning methods? Participants will have to lie on the examination bed while investigator making measurements 7 times in a row on one single location.

DETAILED DESCRIPTION:
Learning effect of MSOT measurements have been observed by previous studies. Therefore, in this study, we aim to quantify the learning effect with circulation-related parameters (Hb, HbO2, SO2) and the similarity between repeated images (structural similarity index measure, SSIM). The measurement would be repeated by 5 different investigators, two of them are professionals, defined as experience over 200 times of MSOT measurement, while the other three are trainees, who haven't performed any MSOT measurements before and each has received one different teaching method, one receiving personal teaching from a professional, one receiving video instruction and one receiving instructions written in paper form.

ELIGIBILITY:
Inclusion Criteria:

-all those who with the age between 18 and 40 year-old

Exclusion Criteria:

* diabetes mellitus
* hypertension
* cardiovascular diseases
* chronic kidney diseases
* amputation in either lower extremities
* tatoos in either lower extremities

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The volunteers would be recruited in the clinic where the research takes place, by posters and public speeches. T
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Learning curve in MSOT measurements. | 5 days
  If the quality of MSOT measurements improved with practices.
Different learning curve between professionals and trainees. | 5 days
  Observe the possible difference between the learning curves in professionals and trainees.

SECONDARY OUTCOMES:
Different learning curve in three different teaching methods | 5 days
  Three trainees, each received different teaching methods, perform the same measurement on the same participants. The outcome is to observe possible difference in learning curve in these three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen-Nuremberg (FAU), Department of Vascular Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No